CLINICAL TRIAL: NCT04124796
Title: Identification of Psychosocial Factors Associated With Diagnostic Delay in Advanced Basal Cell Carcinoma
Acronym: PSYCHO-CBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bordeaux Population Health Research centre (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2018/16
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Basal Cell, Malignant
Keywords: Carcinoma, Basal Cell; psycho-social factors
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Intervention Model Description: * Fifteen to twenty "target subjects" patients are expected, corresponding to the average population received each year for a CBCa in the unit.
  * Fifteen members of the health care team managing these patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- target subjects (Experimental): "target subjects" patients are expected, corresponding to the average population received each year for a CBCa in the unit.
  Interventions: Other: Semi-structured interviews
- health care team (Active Comparator): the health care team managing these patients
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Semi-structured interviews — Based on an interview grid previously built, the interviews will investigate the factors governing the decision to consult and methods of intervention to reduce the time to consult.

SUMMARY:
The aim of this study was to identify psycho-social factors associated with diagnostic delay in advanced basal cell carcinomas. Thus, the objective is to develop recommendations to better identify CBCa populations at risk, improve earlier their diagnosis and thus their care with an adequate and targeted information.

DETAILED DESCRIPTION:
Skin cancers incidence is constantly increasing as a result of ageing of the population, and is then a critical issue of concern. Among skin cancers, basal cell carcinoma is the most common. Its treatment is mainly based on surgery that has to be done early. Indeed, CBC can lead to progressive destruction of tissues and significant morbidity in advanced stages. In these advanced stages (CBCa), they are no longer accessible to surgery or radiation therapy. The recently developed targeted therapies represent a significant therapeutic progress. To date, there are few data -none in France- concerning the cause of diagnostic delay .

Thus, the main goal of this study will be to evidence the brakes and facilitators who chair the decision-making to consult in patients with a CBCa, by investigating:

* the perception of the target subjects (patients);
* the perception of the healthcare team; We will also conduct a critical meta-synthesis (qualitative meta-analysis) of the literature concerning the diagnostic delay and decision-making in onco-dermatology.

It is a prospective non-Interventional exploratory qualitative study without direct individual benefit

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with a CBCa supported for less than 12 months in the onco-Dermatology unit of the CHU de Bordeaux.
* Are defined as locally advanced,tumors with major invasion of adjacent structures, that are not accessible for surgical resection or radiotherapy, .
* Patients will sign a consent after reading the fact sheet explaining the objectives of the study.

Exclusion Criteria:

* subjects with severe dementia (mini mental state less than 10)
* An anonymized list of non-included according to this criterion will be carried out in order to quantify the number of advanced CBC with severe dementia and also the number of refusals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Proportion of "psycho-social factors" that chair the decision-making to consul | Day 1
  semi-structured interviews of patients by the psychologist

CONTACTS AND LOCATIONS:
Overall Officials: Marie BEYLOT BARRY, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Service de Dermatologie - Hôpital Saint André, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garrouteigt C, Broc G, Legrand A, Quintard B, Beylot-Barry M. Facilitators of and obstacles to consultation in patients with advanced basal cell carcinoma: a French pilot study. Arch Dermatol Res. 2021 Dec;313(10):829-835. doi: 10.1007/s00403-020-02175-x. Epub 2021 Jan 12. PMID 33433714